CLINICAL TRIAL: NCT06748469
Title: Analgesic Efficacy of Different Pulse Radiofrequency Treatment Durations in the Management of Lumbosacral Radicular Pain
Brief Title: Efficacy of Pulse Radiofrequency Durations in Lumbosacral Pain
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gülçin Babaoğlu, Medical doctor, Ankara City Hospital Bilkent
Other Study IDs: TABED 1-24-764
Record Dates: First submitted 2024-12-18; First posted 2024-12-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-02

CONDITIONS: RADICULAR PAIN
Keywords: RADICULAR PAIN; DORSAL ROOT GANGLIA; PULSED RADIOFREQUENCY

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with lumbosacral radicular pain: patients with lumbosacral radicular pain resistant to conservative treatments
  Interventions: Procedure: The duration of the intervention will be 240 seconds; Procedure: Dorsal Root Ganglion pulsed radiofrequency 480sec

INTERVENTIONS:
Procedure: The duration of the intervention will be 240 seconds — Dorsal Root Ganglion pulsed radiofrequency 240sec
Procedure: Dorsal Root Ganglion pulsed radiofrequency 480sec — The duration of the intervention will be 480 seconds

SUMMARY:
Brief Summary:

This study aims to compare the efficacy of short-duration (240 sec) and long-duration (480 sec) pulsed radiofrequency (PRF) applications on pain, functionality, patient satisfaction, and side effect profiles in patients with lumbosacral radicular pain. The PRF procedure will be applied to the dorsal root ganglion (DRG) under fluoroscopic guidance.

DETAILED DESCRIPTION:
In this study, all procedures will be performed in the prone position under sterile conditions and guided by fluoroscopy. After identifying anatomical landmarks, the cannula will be positioned close to the dorsal root ganglion. The tip of the cannula will be placed in the dorsal-cranial quadrant of the intervertebral foramen in the lateral view, and between one-third and halfway along the pedicle column in the anteroposterior view. Once the RF cannula is properly positioned, an RF electrode will be inserted through the cannula and connected to the RF generator. The final position of the RF cannula will be confirmed by sensory stimulation (paresthesia) at less than 0.5 V and motor stimulation perceived at a level at least 1.5 times greater than the sensory stimulation threshold.

In the short-duration PRF group, a PRF cycle will be applied at 42°C for 240 seconds, while in the long-duration group, it will be applied at 42°C for 480 seconds. Following the PRF application, epidural spread will be confirmed using contrast dye, after which 4 mL of a solution containing 8 mg dexamethasone and 5 mg bupivacaine will be injected at each level.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Pain severity NRS ≥ 4
* Pain duration > 12 weeks Refractory to conservative treatments (physical therapy, medical treatments) Exclusion Criteria Malignancy-related pain Diagnosis of diabetes mellitus or polyneuropathy Back pain more severe than leg pain Conditions that impair follow-up (e.g., psychiatric disorders, dementia) Patients refusing the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to undergo DRG PRF for lumbar radicular pain in bilkent city hospital algology clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale on pain severity (0 = no pain, 10 = unbearable pain)) | 1, 3, and 6 months
  Change in pain severity

SECONDARY OUTCOMES:
Global perceived effect (GPE) | 1, 3, and 6 months
  Change in GPE scores according to the 7-point Likert scale (1=worst, 7=best) over time will be used to assess patient satisfaction and improvement
Oswetry disability index (ODI) | 0, 1, 3, and 6 months
  Change in 10-item Oswestry disability index (ODI) questionnaire (range: 0-100; 0 = no disablility) over time will be used to assess physical function
Patient satisfaction | 1, 3, and 6 months
  Change in Patient satisfaction (5-point Likert scale, 0= very disappointed, 5=very satisfied) over time will be used
Change in analgesic use | 1, 3, and 6 months
  Change in analgesic use over time (0=same, 1=decreased, 2=increased)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Pain Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ı don't want

REFERENCES:
- [Result] Wan C, Dong DS, Song T. High-Voltage, Long-Duration Pulsed Radiofrequency on Gasserian Ganglion Improves Acute/Subacute Zoster-Related Trigeminal Neuralgia: A Randomized, Double-Blinded, Controlled Trial. Pain Physician. 2019 Jul;22(4):361-368. PMID 31337167
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31337167/